CLINICAL TRIAL: NCT01058967
Title: UTHSC-H Proposal for Prospective Evaluation of Aeromedical EMS Ultrasound in Major Trauma Victims.
Brief Title: Prospective Evaluation of Aeromedical EMS Ultrasound in Major Trauma Victims
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: SonoSite, Inc. (Industry)
Responsible Party: Principal Investigator, Sara K Miller, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-08-0085
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Major Trauma Patients
Keywords: Code III trauma (highest acuity); Life Flight aeromedical ambulance service

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- major trauma victims: Code 3 patients (highest acuity) admitted to hospital via air ambulance service

SUMMARY:
The purpose of this study is to investigate the use of ultrasound by aeromedical prehospital providers.

DETAILED DESCRIPTION:
This study will be divided into three parts. The first portion involves the education/inservices of the aeromedical prehospital providers to document the knowledge and skills necessary to perform and interpret eFAST exams using ultrasound pre hospitalization.

The second portion involves testing the logistics of utilization of prehospital ultrasound. Data will be collected by the participating aeromedical prehospital providers to rate the durability of the equipment, difficulty in preforming the eFAST exam, interference with other actions and ability of retention of images.

The third portion will involve the aeromedical prehospital providers performing the eFAST exam using the ultrasound prehospital and comparing their findings with the gold standard exam, CT scan, while patient is in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Code 3 trauma activation Admitted directly from scene Transported via Life Flight (aeromedical ambulance)

Exclusion Criteria:

* transfer from outside hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have experienced a major traumatic injury highest acuity trauma activation (Code III status) transported from scene to hospital via Life Flight (hospital aeroambulance service)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this study is to determine if the aeromedical prehospital providers are able to accurately and rapidly perform and interpret eFAST exams in major trauma victims. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Greg Press, MD, Principal Investigator — UTHSC-Houston
Locations (1):
- Memorial Hermann Hospital - Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Press GM, Miller SK, Hassan IA, Alade KH, Camp E, Junco DD, Holcomb JB. Prospective evaluation of prehospital trauma ultrasound during aeromedical transport. J Emerg Med. 2014 Dec;47(6):638-45. doi: 10.1016/j.jemermed.2014.07.056. Epub 2014 Oct 1. PMID 25281177